CLINICAL TRIAL: NCT02202174
Title: The Safety and Efficacy of Supraglottic Airway Use in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Narasimhan Jagannathan, Primary Investigator; MD, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2014-15832
Record Dates: First submitted 2014-07-25; First posted 2014-07-28 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Supraglottic Airway Use in Children
Keywords: supraglottic airway; children; safety; efficacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Supraglottic Airway Device: Patients will receive a supraglottic airway device as a primary means of ventilation. The following devices may be used: LMA Unique, LMA ProSeal, LMA Supreme, LMA Flexible, Ambu Aura-I, Ambu Aura Once, Air-Q, I-Gel, or other supraglottic airway device. Choice of the device will be clinician dependent and based on the patients body weight per manufacturer guidelines
  Interventions: Device: Supraglottic Airway Device

INTERVENTIONS:
Device: Supraglottic Airway Device
  Other Names: LMA Unique; LMA ProSeal; LMA Supreme; LMA Flexible; Ambu Aura-i; Ambu Aura Once; Air-Q; I-Gel

SUMMARY:
This purpose of this study is to determine the effectiveness, risk factors, and complications associated with use of supraglottic airway devices for primary airway maintenance during routine anesthesia in children.

DETAILED DESCRIPTION:
This study aims to understand the efficacy of supraglottic airway (SGA) use in children in a tertiary care Children's Hospital.

Observational data regarding the type of SGA, experience level of practitioner, placement technique, number of placement attempts or placement failure, device failure, and cause of any related peri-operative complications will be prospectively collected.

The data collected in this study will allow the investigators to assess the overall safety and efficacy of SGA use in various medical and surgical procedures performed under general anesthesia in children.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing anesthesia with use of a supraglottic airway device as a primary means of oxygenation & ventilation

Exclusion Criteria:

* N/A

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients undergoing anesthesia with use of a supraglottic airway device as primary means of oxygenation and ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Supraglottic Airway Device Failure | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Occurrence and reason for supraglottic airway device failure (ie inadequate ventilation, laryngospasm, bronchospasm, etc) will be recorded in addition to conversion to tracheal intubation

SECONDARY OUTCOMES:
Ease of Placement of Supraglottic Airway Device | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Ease of placement of supraglottic airway device ranging from 1 (easy) to 4 (difficult)
Multiple Attempts to Place Supraglottic Airway Device | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  change in device, placement method, and provider will be recorded
Airway Maneuvers/interventions | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  the number and type of airway maneuvers performed after device placement and during maintenance will be recorded
Occurrence of Inadequate Ventilation | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  cause and solution for inadequate ventilation will be recorded
Intraoperative Complications | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Time period of complication (ie during device placement, maintenance, or removal) and cause of complication (ie. dental injury, light anesthesia, regurgitation, laryngospasm, bronchospasm, aspiration, etc.) will be recorded
Postoperative Complications | participants will be followed for the duration of anesthesia and 24 hours postoperatively
  Complications noted postoperatively relating to reflex activation of the airway, sore throat, or hoarseness

CONTACTS AND LOCATIONS:
Overall Officials: Narasimhan Jagannathan, MD, Principal Investigator — Ann & Robert H. Lurie Children's Hospital of Chicago / Stanley Manne Research Institute
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Jagannathan N, Sequera-Ramos L, Sohn L, Wallis B, Shertzer A, Schaldenbrand K. Elective use of supraglottic airway devices for primary airway management in children with difficult airways. Br J Anaesth. 2014 Apr;112(4):742-8. doi: 10.1093/bja/aet411. Epub 2013 Dec 8. PMID 24322570
- [Background] Asai T. Is it safe to use supraglottic airway in children with difficult airways? Br J Anaesth. 2014 Apr;112(4):620-2. doi: 10.1093/bja/aeu005. Epub 2014 Feb 20. No abstract available. PMID 24561643
- [Background] Lopez-Gil M, Brimacombe J, Alvarez M. Safety and efficacy of the laryngeal mask airway. A prospective survey of 1400 children. Anaesthesia. 1996 Oct;51(10):969-72. doi: 10.1111/j.1365-2044.1996.tb14968.x. PMID 8984875
- [Background] Bordet F, Allaouchiche B, Lansiaux S, Combet S, Pouyau A, Taylor P, Bonnard C, Chassard D. Risk factors for airway complications during general anaesthesia in paediatric patients. Paediatr Anaesth. 2002 Nov;12(9):762-9. doi: 10.1046/j.1460-9592.2002.00987.x. PMID 12519134
- [Background] Lalwani K, Richins S, Aliason I, Milczuk H, Fu R. The laryngeal mask airway for pediatric adenotonsillectomy: predictors of failure and complications. Int J Pediatr Otorhinolaryngol. 2013 Jan;77(1):25-8. doi: 10.1016/j.ijporl.2012.09.021. Epub 2012 Oct 11. PMID 23063385
- [Background] Mathis MR, Haydar B, Taylor EL, Morris M, Malviya SV, Christensen RE, Ramachandran SK, Kheterpal S. Failure of the Laryngeal Mask Airway Unique and Classic in the pediatric surgical patient: a study of clinical predictors and outcomes. Anesthesiology. 2013 Dec;119(6):1284-95. doi: 10.1097/ALN.0000000000000015. PMID 24126262